CLINICAL TRIAL: NCT05798481
Title: A Pilot Pre-Phase 1 Clinical Trial to Study How Administering Sublingual Nitric Oxide Donor S-nitroso-N-acetylcysteine Affects the Systemic Blood Pressure in Healthy Human Volunteers.
Brief Title: Effect of Sublingually Generated S-nitroso-N-acetylcysteine on Systemic Blood Pressure.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nagababu Enika, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300010325
Record Dates: First submitted 2023-03-10; First posted 2023-04-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Nitric oxide; Sodium nitrite; N-acetylcysteine; S-nitrosothiols; systemic blood pressure; Vasodilators; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: The optimum levels of 2.5 mg and 5mg mg sodium nitrite and fixed amount of 50 mg N-acetylcysteine are used for this study. Total of 14 subjects are divided to two groups.Group 1 is tested with the low dose of 2.5 mg sodium nitrite. If no adverse effects are noticed in this group, the study is proceed for 2nd group with 5mg sodium nitrite.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- sodium nitrite and N-acetycysteine mixture (Experimental): sodium nitrite 2.5mg + N-acetylcysteine 50mg
  Sodium nitrite 5 mg + N-acetylcysteine 50mg
  Interventions: Drug: Mixture of Sodium Nitrite and N-acetylcysteine (NAC) crytals.

INTERVENTIONS:
Drug: Mixture of Sodium Nitrite and N-acetylcysteine (NAC) crytals. — Exactly 2.5 mg or 5 mg sodium nitrite and 50 mg N-acetylcysteine are weighed and mixed together just before use. The mixture is placed under the participant's tongue. The powder slowly dissolves in saliva and generate S-nitrosoacetylcysteine. Investigators will ask the subjects not to swallow the drug at least for 30 min. Administration of nitrite and N-acetylcysteine individually at these concentrations is not expected to change any blood NO chemistry or the systemic blood pressure. Hence, investigators will not investigate the effects of nitrite and N-acetylcysteine individually in this study. Placebo control is not needed for this study because the baseline parameters will serve as control. Investigators will assess the drug effect based on the difference between pre-treatment and post-treatment values.

SUMMARY:
The purpose of the study is to increase the in vivo levels of nitric oxide by generating nitric oxide donor compound S-nitrosoacetylcysteine (SNOAC) using the mixture of sodium nitrite and N-acetylcysteine crystals in the sublingual space. The generated SNOAC rapidly diffuses into blood circulation thereby decrease the systemic blood pressure. This compound can be an alternative to organic nitrate NO donor drugs without developing tolerance in patients.

DETAILED DESCRIPTION:
It is well established that increasing the bioavailability of endogenous nitric oxide (NO) protects against cardiovascular diseases. Administering exogenous NO donors is one option to increase endogenous NO levels. Organic nitrates like nitroglycerin have been used as NO donors to protect against angina and ischemic heart failure for over a century. However, their therapeutic value is compromised by rapid development of tolerance during sustained therapy. Hence, these drugs cannot be used as sustain sources of NO. Low-molecular-weight S-nitrosothiols are proven NO donors that have potent vasodilatory, antithrombotic, and anti-inflammatory activities. However, their prophylactic use is hindered by instability after preparation. Inorganic nitrite is emerging as a hypoxic vasodilator, but recent clinical studies indicate that high oral doses of >100 mg/day are required to improve vascular tone. To solve the problems of organic nitrates tolerance, S-nitrosothiol instability, and high nitrite dose requirements, the technique of generating S-nitrosoacetylcysteine (SNOAC) sublingually or in the stomach by reacting sodium nitrite with N-acetylcysteine (NAC) in rodent models was developed. This SNOAC is rapidly absorbed into circulation and increases plasma S-nitrosothiols and reduces systemic systolic and diastolic blood pressure. The major objective of the proposed pre-phase 1 study is to confirm the preclinical findings, including whether the procedure used to generate and deliver NO is feasible in humans using optimal levels of nitrite (2.5mg and 5mg) and NAC (50mg) and a minimum number of subjects. The study will assess the feasibility of using nitrite and NAC mixture sublingually, generation and absorption of SNOAC into circulation, and blood pressure response to the optimum doses of nitrite and NAC. This study will lay the groundwork for determining whether this NO delivery technique can be implemented to initiate comprehensive clinical studies. S-nitrosothiols, nitrite, and nitrate in plasma will be measured by highly sensitive chemiluminescence assay and monitor cardiovascular hemodynamics by FDA-approved mobil-O-graph for ambulatory subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects who are at least 21 years old and who consent to participate in the study.
* Participants must be willing to have approximately 15 mL of blood drawn via venipuncture and undergo blood pressure measurement.

Exclusion Criteria:

* Individuals who are below 21 years of age, pregnant, have major cardiovascular problems or sickle cell disease, incarcerated individuals or are unable to give consent will be excluded.
* Those whose blood pressure is below normal (i.e., 120/80) and those who have cardiovascular problems and taking organic nitrates and sildenafil-based drugs will also be excluded.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
Measurement of plasma nitrite, nitrate and S-nitrosothiols in the study participants. | up to 18 months
  Plasma level of nitrite, nitrate and S-nitrosothiols species (nanomol/L) will be measured by highly validated ozone-based chemiluminescience assay before, during and the end of sublingual administration of S-nitrosoacetylcysteine in study participants The drug effect will be assessed based on the change in the nitrite, nitrate and S-nitrosothiol values from the baseline levels following the administration of the drug.
Measurement of Systemic systolic and diastolic blood pressure | up to 11 months
  The FDA approved Mobil-O-Graph blood pressure (BP) apparatus will be used to measure the BP parameters. BP is measured in units of millimeters of mercury (mmHg). The cuff will be wrapped around the left arm and the measurement time will be set for 120 minutes. Blood pressure parameters will be automatically measured at 2-minute intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nagababu Enika, PhD, Principal Investigator — University of Alabama at Birmingham; Brant Wagener, MD, PhD, Study Director — University of Alabama at Birmingham
Locations (1):
- Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All the data will be shared through abstracts, presentation at conferences and publications.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: August 2024
Access Criteria: www.clinicaltrials.gov and UAB websites

REFERENCES:
- [Background] Farah C, Michel LYM, Balligand JL. Nitric oxide signalling in cardiovascular health and disease. Nat Rev Cardiol. 2018 May;15(5):292-316. doi: 10.1038/nrcardio.2017.224. Epub 2018 Feb 1. PMID 29388567
- [Background] Secker-Walker LM, Craig JM, Hawkins JM, Hoffbrand AV. Philadelphia positive acute lymphoblastic leukemia in adults: age distribution, BCR breakpoint and prognostic significance. Leukemia. 1991 Mar;5(3):196-9. PMID 2013979
- [Background] Munzel T, Daiber A, Gori T. More answers to the still unresolved question of nitrate tolerance. Eur Heart J. 2013 Sep;34(34):2666-73. doi: 10.1093/eurheartj/eht249. Epub 2013 Jul 17. PMID 23864131
- [Background] Al-Sa'doni H, Ferro A. S-Nitrosothiols: a class of nitric oxide-donor drugs. Clin Sci (Lond). 2000 May;98(5):507-20. PMID 10781381
- [Background] Sun J, Murphy E. Protein S-nitrosylation and cardioprotection. Circ Res. 2010 Feb 5;106(2):285-96. doi: 10.1161/CIRCRESAHA.109.209452. PMID 20133913
- [Background] Daiber A, Xia N, Steven S, Oelze M, Hanf A, Kroller-Schon S, Munzel T, Li H. New Therapeutic Implications of Endothelial Nitric Oxide Synthase (eNOS) Function/Dysfunction in Cardiovascular Disease. Int J Mol Sci. 2019 Jan 7;20(1):187. doi: 10.3390/ijms20010187. PMID 30621010